CLINICAL TRIAL: NCT02411968
Title: Follow up After Percutaneous MR-guided Cryoablation of Small Renal Masses.
Brief Title: Follow up After Cryoablation of Small Renal Masses.
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL48292.091.14
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: Cryosurgery; Carcinoma, renal cell; Diagnostic Imaging; Diagnostic techniques, urological; Radionuclide imaging; Follow up
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Needle biopsy kidney tumor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 111In-Girentuximab DOTA SPECT: Patients >50 years of age with renal tumours ≤4 cm highly suspicious for a malignancy planned to undergo cryotherapy will undergo 111In-Girentuximab DOTA SPECT scanning.
  Interventions: Other: 111In-Girentuximab DOTA SPECT

INTERVENTIONS:
Other: 111In-Girentuximab DOTA SPECT

SUMMARY:
Currently there is no consensus on post procedural follow up imaging following percutaneous cryoablation of renal tumors. Interpretation of conventional contrast enhanced imaging (CT and MRI) during follow up can be very challenging. The objective of this study is to evaluate the feasibility of early evaluation of the therapeutic effect by performing early follow up imaging after percutaneous MR-guided cryoablation of pT1a renal cell carcinoma using 111In-Girentuximab-DOTA SPECT CT imaging.

DETAILED DESCRIPTION:
With the growing number of small renal masses (SRMs) detected, a growing interest in minimal invasive treatment options for these lesions is seen as they come with several advantages compared to partial nephrectomy. Current guidelines state that patients with a small renal mass unfit to undergo surgery, should be considered for minimal invasive ablative treatment. Although percutaneous cryoablation is shown to be a safe and effective therapy for SRM, there is no consensus on post procedural follow up imaging which should be aimed at evaluation of therapeutic effect of the intervention and the early detection of residual and recurrent disease. Also interpretation of conventional contrast enhanced imaging (CT and MRI) during follow up can be very challenging due to contrast enhancement not necessarily indicating residual or recurrent disease.

The objective of this study is to evaluate the feasibility of early evaluation of the therapeutic effect by performing early follow up imaging after percutaneous MR-guided cryoablation of pT1a renal cell carcinoma 111In-Girentuximab-DOTA SPECT CT imaging.

Therefore, before cryoablation, a targeting 111In-Girentuximab-DOTA SPECT CT scan is performed. Additional functional 111In-Girentuximab-DOTA SPECT CT scan 4-6 weeks after percutaneous MR-guided cryoablation of small renal masses is performed. The latter will take place in case of proven targeting on the pre procedural 111In-Girentuximab-DOTA SPECT CT scan. Standard 1 and 3 months follow up MRI after treatment is performed.

ELIGIBILITY:
Inclusion Criteria:

* >50 years of age;
* At least one untreated T1a tumour of one kidney (tumour ≤ 4 cm in greatest dimension);
* Signed IRB-approved informed consent form.

Exclusion Criteria:

* Pregnancy or breast feeding;
* Known hypersensitivity or HACA against Girentuximab.
* Administration of experimental medication for imaging purposes within three months before administration of Indium-111-Girentuximab for this study, except the administration of Girentuximab labeled with a random isotope.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >50 years of age with renal tumours ≤4 cm highly suspicious for a malignancy on imaging requiring treatment and planned to undergo cryotherapy.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Predictive value. | Up to at least 3 months following initial treatment (cryoablation).
  Positive predictive value and negative predictive value of 111In-Girentuximab-DOTA SPECT 4-6 weeks after intervention as confirmed on subsequent conventional follow up imaging (contrast enhanced MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen J Futterer, M.D. PhD, Principal Investigator — Radboud University Medical Center; Wim JG Oyen, M.D. PhD, Principal Investigator — Radboud University Medical Center; Peter FA Mulders, M.D. PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No